CLINICAL TRIAL: NCT01831310
Title: Effects Of Standard And/Or Glutamine Dipeptide And/Or Omega-3 Fatty Ascid-Supplemented Parenteral Nutrition On Neutrophil Functions, Interleukin-8 Level And Length Of Stay-A Double Blind,Controlled, Randomized Study
Brief Title: Nutrition for Colorectal Cancer Patients and Neutrophil Functions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Nuh Zafer Cantürk, Professor in Surgical Oncology and head of Nutrition Team, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Canturkz1; KOUNutrition1 (Other: Kocaeli University)
Record Dates: First submitted 2013-04-01; First posted 2013-04-15 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Malnutrition; Colorectal Cancer
Keywords: Colorectal cancer; nutrition; neutrophil phagocytosis; neutrophil adhesivity; glutamine; omega 3 fatty acids
MeSH Terms: conditions — Malnutrition; Colorectal Neoplasms | interventions — alanylglutamine; fish oil triglycerides

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (standard) (Kabiven) (Active Comparator): an isocaloric and iso-nitrogenous standard parenteral nutrition (Kabiven)
  Interventions: Dietary Supplement: Standard (Kabiven)
- Standard parenteral-glutamine (S-D) (Experimental): alanine-glutamine (aln-gln) (Dipeptiven) supplemented parenteral nutrition (S-D group, n=8),
  Interventions: Dietary Supplement: Standard-Glutamine
- Standard-Omega-3 fatty acid (S-O) (Experimental): Omega-3 fatty acid (Omegaven) supplemented parenteral nutrition (S-O group, n=8)
  Interventions: Dietary Supplement: Standard-Omega 3 fatty acid
- Standard-glutamine-omega 3 (S-D-O) (Experimental): ala-gln and omega 3 fatty ascid supplemented parenteral nutrition (S-D-O group, n=10).
  Interventions: Dietary Supplement: Standard-glutamine-omega 3

INTERVENTIONS:
Dietary Supplement: Standard (Kabiven) — Parenteral nutrition provided 25-30 kcal/kg/day energy and 0.15-0.20 g/kg/day nitrogen. All nutrient substrates were mixed in 3 litre bags and infused in 24 h through a dedicated central venous line
  Arms: Control (standard) (Kabiven)
Dietary Supplement: Standard-Glutamine — Parenteral nutrition (Kabiven) provided 25-30 kcal/kg/day energy and 0.15-0.20 g/kg/day nitrogen. it was 0.3-0.4 g/kg/day for glutamine dipeptide (Dipeptiven) supplementation. All nutrient substrates were mixed in 3 litre bags and infused in 24 h through a dedicated central venous line
  Other Names: Standard (Kabiven)-Glutamine (Dipeptiven)
  Arms: Standard parenteral-glutamine (S-D)
Dietary Supplement: Standard-Omega 3 fatty acid — Parenteral nutrition (Kabiven) provided 25-30 kcal/kg/day energy and 0.15-0.20 g/kg/day nitrogen. The dose of omega 3 fatty acid (omegaven)supplementation was 0.1-0.2 g/kg /day. All nutrient substrates were mixed in 3 litre bags and infused in 24 h through a dedicated central venous line
  Other Names: Standard (Kabiven)-Omega 3 fatty acid(Omegaven)
  Arms: Standard-Omega-3 fatty acid (S-O)
Dietary Supplement: Standard-glutamine-omega 3 — Parenteral nutrition (kabiven) provided 25-30 kcal/kg/day energy and 0.15-0.20 g/kg/day nitrogen. The dose of omega 3 fatty acid (omegaven) supplementation was 0.1-0.2 g/kg /day and it was 0.3-0.4 g/kg/day for glutamine dipeptide (dipeptiven)supplementation. All nutrient substrates were mixed in 3 litre bags and infused in 24 h through a dedicated central venous line
  Other Names: Standard (Kabiven)-glutamine (Dipeptiven)-omega 3 (Omegaven)
  Arms: Standard-glutamine-omega 3 (S-D-O)

SUMMARY:
Hypercatabolism and immune suppression are frequently seen in patients with malignancy. Preoperative nutritional state is an important factor in determining surgical and postoperative complications because the preoperative nutritional status affects the postoperative nutritional state, immunity and inflammatory response. In these patients, standard parenteral nutrition may not be sufficient to maintain the immunity and provide positive or stabilized nitrogen balance. Preoperative and perioperative supplementation with immune-enhancing enteral nutrition has been reported to increase total lymphocytes and T lymphocytes and decrease circulating levels of interleukin 6 and tumor necrosis factor- alfa. There is a report which showed that glutamine dipeptide supplemented parenteral nutrition improved the cellular and humoral immune functions. The investigators aimed to evaluate the effect of postoperative glutamine-dipeptide and/or omega 3 fatty acid supplemented parenteral nutrition on the neutrophil functions and postoperative course of patients with colorectal cancer.

DETAILED DESCRIPTION:
Purpose Hypercatabolism and immune suppression are frequently seen in patients with malignancy.Preoperative nutritional state is an important factor in determining surgical and postoperative complications because the preoperative nutritional status affects the postoperative nutritional state, immunity and inflammatory response.In these patients, standard parenteral nutrition may not be sufficient to maintain the immunity and provide positive or stabilized nitrogen balance. Preoperative and perioperative supplementation with immune-enhancing enteral nutrition has been reported to increase total lymphocytes and T lymphocytes and decrease circulating levels of interleukin 6 and tumor necrosis factor- alfa.There is a report which showed that glutamine dipeptide supplemented parenteral nutrition improved the cellular and humoral immune functions. The investigators aimed to evaluate the effect of postoperative glutamine-dipeptide and/or omega 3 fatty acid supplemented parenteral nutrition on the neutrophil functions and postoperative course of patients with colorectal cancer.

Condition Intervention Phase Malnutrition Colorectal Cancer Dietary Supplement: Immunonutrition Phase 4

Study Type: Interventional Study Design: Prevention, Parallel Assignment, Double Blind (Subject, Investigator), Randomized, N/A

Official Title: Effects Of Standard And/Or Glutamine Dipeptide And/Or Omega-3 Fatty Ascid-Supplemented Parenteral Nutrition On Neutrophil Functions, Interleukin-8 Level And Length Of Stay-A Double Blind,Controlled, Randomized Study

Primary Outcome Measure: Title: neutrophil functions Time Frame: perioperative,postoperative third and seventh days for change in first seven days of hospital stay Description: For comparison of four different nutrition on neutrophil functions in first seven days of hospital stays.

Secondary Outcome Measures: Title: Length of stay Time Frame: Length of stay (participants will be followed for the duration of hospital stay) for colorectal cancer patients which are eligable for study study from january 2007 to january 2008 in one year period.

Description: For comparison of four different nutrition on length of stay (participants will be followed for the duration of hospital stay)

Actual Enrollment: 36 Study Start Date: January 2007 Actual Study Completion Date: January 2008 Actual Primary Completion Date: January 2008

Arms Assigned Interventions Active Comparator: Control an isocaloric and iso-nitrogenous standard parenteral nutrition

Dietary Supplement: Immunonutrition Parenteral nutrition provided 25-30 kcal/kg/day energy and 0.15-0.20 g/kg/day nitrogen. The dose of omega 3 fatty acid supplementation was 0.1-0.2 g/kg /day and it was 0.3-0.4 g/kg/day for glutamine dipeptide supplementation. All nutrient substrates were mixed in 3 litre bags and infused in 24 h through a dedicated central venous line

Experimental: Standard parenteral-glutamine (S-D) alanine-glutamine (aln-gln) (Dipeptiven) supplemented parenteral nutrition (S-D group, n=8),

Dietary Supplement: Immunonutrition Parenteral nutrition provided 25-30 kcal/kg/day energy and 0.15-0.20 g/kg/day nitrogen. The dose of omega 3 fatty acid supplementation was 0.1-0.2 g/kg /day and it was 0.3-0.4 g/kg/day for glutamine dipeptide supplementation. All nutrient substrates were mixed in 3 litre bags and infused in 24 h through a dedicated central venous line

Experimental: Standard-Omega-3 fatty acid (S-O) Omega-3 fatty acid (Omegaven) supplemented parenteral nutrition (S-O group, n=8)

Dietary Supplement: Immunonutrition Parenteral nutrition provided 25-30 kcal/kg/day energy and 0.15-0.20 g/kg/day nitrogen. The dose of omega 3 fatty acid supplementation was 0.1-0.2 g/kg /day and it was 0.3-0.4 g/kg/day for glutamine dipeptide supplementation. All nutrient substrates were mixed in 3 litre bags and infused in 24 h through a dedicated central venous line

Experimental: Standard-glutamine-omega 3 (S-D-O) ala-gln and omega 3 fatty ascid supplemented parenteral nutrition (S-D-O group, n=10).

Dietary Supplement: Immunonutrition Parenteral nutrition provided 25-30 kcal/kg/day energy and 0.15-0.20 g/kg/day nitrogen. The dose of omega 3 fatty acid supplementation was 0.1-0.2 g/kg /day and it was 0.3-0.4 g/kg/day for glutamine dipeptide supplementation. All nutrient substrates were mixed in 3 litre bags and infused in 24 h through a dedicated central venous line

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer patients who were included study were between 50 and 70 years old

Exclusion Criteria:

* preoperatively suffered from serious comorbid chronic disease and received chemotherapy and radiotherapy
* immunosuppressive and /or immunomodulator drugs in last 6 months

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
neutrophil functions | perioperative,postoperative third and seventh days for change in first seven days of hospital stay
  For comparison of four different nutrition on neutrophil functions in first seven days of hospital stays.

SECONDARY OUTCOMES:
Length of stay | Length of stay (participants will be followed for the duration of hospital stay) for colorectal cancer patients which are eligable for study study from january 2007 to january 2008 in one year period.
  For comparison of four different nutrition on length of stay (participants will be followed for the duration of hospital stay)

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Dulger, Professor, Study Chair — Kocaeli University
Locations (1):
- Kocaeli University School of Medicine, Kocaeli, Turkey (Türkiye)